CLINICAL TRIAL: NCT06626607
Title: A Study of the Effect of Different Antihypertensive Drugs on the Disease Progression of Aortic Dissection/Aneurysm
Brief Title: Different Antihypertensive Drugs on Aortic Diseases
Acronym: DADAD
Status: Completed | Type: Observational
Sponsor: Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Zhang Tingting, Professor, Eighth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: ZB-KYIRB-AF/SC-08/02.0
Record Dates: First submitted 2024-09-30; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Aortic Aneurysm; Aortic Dissection
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CCB group: Patients' postoperative antihypertensive includes CCB (Calcium Calcium Entry Blockers)
  Interventions: Drug: CCB use
- non-CCB group: Patients' postoperative antihypertensive does not include CCB
  Interventions: Drug: non-CCB use

INTERVENTIONS:
Drug: CCB use — Postoperative antihypertensive medication includes CCB
  Groups: CCB group
Drug: non-CCB use — Postoperative antihypertensive medication does not include CCB
  Groups: non-CCB group

SUMMARY:
The goal of this observational study is to learn about the effect of different hypotensive drugs on the prognosis of postoperative aortic patients. The main question it aims to answer is:

Does different hypotensive drugs influence the prognosis of postoperative aortic patients? As participants already taking hypotensive drugs as part of their regular medical care, the investigators collect the participants' pre-operation medical record and post-operative follow-up record to evaluate the aorta condition.

DETAILED DESCRIPTION:
This study is a cohort study that aims to explore the effects of different antihypertensive regimens on aortic remodelling in patients after aortic surgery by collecting the hospitalization and outpatient follow-up data. The study plans to gather perioperative and postoperative follow-up data from over 600 patients who underwent aortic surgery at the Eighth Affiliated Hospital and Beijing Anzhen Cardiothoracic Surgery Center. Patients were assigned based on the postoperative antihypertensive medication regimens. Datas was collected to compare the cardiovascular-related prognoses.

This study primarily includes patients who take oral antihypertensive medications after aortic surgery. The main observations will focus on postoperative complications related to the aorta (such as death, reoperation, dilation, etc.) and aortic diameters after the administration of different antihypertensive medications. Multivariate regression analysis will be employed to investigate the impact of different antihypertensive regimens on patients after aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

* aortic diseases' patients underwent aortic surgery who require antihypertensive medication.

Exclusion Criteria:

* Patients with active vasculitis;
* Patients allergic to contrast agent
* Patients with aorta variation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 1, 2017 to December 1, 2023, 704 patients with hypertention underwent aortic surgery in the institutions. These patients have complete medical records and follow-up data.
Sampling Method: Non-Probability Sample
Enrollment: 704 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Aortic diameter | Through the study completion, on an average of 3 years
  The maximum diameter of the aorta measured by computed tomography angiography

SECONDARY OUTCOMES:
Number of Participants with adverse aortic event | Through the study completion, on an average of 3 years
  Postoperative adverse aortic event during follow-up, including aortic related death or reoperation

IPD SHARING:
Plan to Share IPD: Undecided
The investigators need to consult with the IRB committee.